CLINICAL TRIAL: NCT02012491
Title: Comparative Effectiveness of Pregnancy Failure Management Regimens
Acronym: PreFaiR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 818434; 1R01HD071920-01A1 (NIH)
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Results first posted 2018-12-21 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Spontaneous Abortion
Keywords: Spontaneous abortion; Early Pregnancy Failure; Mifepristone; Misoprostol
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Misoprostol; Mifepristone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- misoprostol plus mifepristone (Active Comparator): 800 micrograms vaginal misoprostol, preceded by 200 milligrams oral mifepristone 24 hours prior
  Interventions: Drug: Misoprostol; Drug: Mifepristone
- misoprostol (Active Comparator): 800 micrograms of vaginal misoprostol alone
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol
  Other Names: Cytotec
Drug: Mifepristone
  Other Names: Mifeprex
  Arms: misoprostol plus mifepristone

SUMMARY:
The purpose of the study is to compare the effectiveness of combination treatment (mifepristone premedication plus single-dose misoprostol) to single-dose misoprostol (standard of care) for the management of early pregnancy failure.

ELIGIBILITY:
Inclusion Criteria:

* between 5 and 12 completed weeks gestation
* 18 years or older
* hemodynamically stable
* confirmed diagnosis of intrauterine embryonic/fetal demise or anembryonic gestation (ultrasound examination demonstrates a fetal pole without cardiac activity measuring between 5.3 and 40 mm or an abnormal growth pattern diagnostic of early pregnancy failure)
* willing and able to give informed consent

Exclusion Criteria:

* diagnosis of incomplete or inevitable abortion (absent gestational sac and/or active bleeding, open cervical os)
* contraindication to mifepristone (chronic corticosteroid administration, adrenal disease)
* contraindication to misoprostol (glaucoma, mitral stenosis, sickle cell anemia, or known allergy to prostaglandin)
* cardiovascular disease (angina, valvular disease, arrhythmia, or cardiac failure)
* most recent hemoglobin <9.5 g/dL
* diagnosis of porphyria
* known clotting defect or receiving anticoagulants
* pregnancy with an intrauterine device (IUD) in place
* breastfeeding during the first 7 days of study participation
* unwilling to comply with the study protocol and visit schedule
* any evidence of viable pregnancy
* possibility of ectopic pregnancy
* known or suspected pelvic infection
* concurrent participation in any other interventional trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-01; Primary Completion 2017-05-15 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney A Schreiber, MD, MPH, Principal Investigator — University of Pennsylvania; Mitchell Creinin, MD, Principal Investigator — University of California, Davis
Locations (3):
- United States (3):
  - University of California, Davis Medical Center, Sacramento, California
  - Montefiore Medical Center, The Bronx, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Nagendra D, Gutman SM, Koelper NC, Loza-Avalos SE, Sonalkar S, Schreiber CA, Harvie HS. Medical management of early pregnancy loss is cost-effective compared with office uterine aspiration. Am J Obstet Gynecol. 2022 Nov;227(5):737.e1-737.e11. doi: 10.1016/j.ajog.2022.06.054. Epub 2022 Jun 30. PMID 35780811
- [Derived] Roe AH, McAllister A, Flynn AN, Martin B, Jiang E, Koelper N, Schreiber CA. The effect of mifepristone pretreatment on bleeding and pain during medical management of early pregnancy loss. Contraception. 2021 Oct;104(4):432-436. doi: 10.1016/j.contraception.2021.04.023. Epub 2021 Apr 28. PMID 33930380
- [Derived] Shorter JM, Koelper N, Sonalkar S, Oquendo MA, Sammel MD, Schreiber CA. Racial Disparities in Mental Health Outcomes Among Women With Early Pregnancy Loss. Obstet Gynecol. 2021 Jan 1;137(1):156-163. doi: 10.1097/AOG.0000000000004212. PMID 33278280
- [Derived] Sonalkar S, Koelper N, Creinin MD, Atrio JM, Sammel MD, McAllister A, Schreiber CA. Management of early pregnancy loss with mifepristone and misoprostol: clinical predictors of treatment success from a randomized trial. Am J Obstet Gynecol. 2020 Oct;223(4):551.e1-551.e7. doi: 10.1016/j.ajog.2020.04.006. Epub 2020 Apr 17. PMID 32305259
- [Derived] Nagendra D, Koelper N, Loza-Avalos SE, Sonalkar S, Chen M, Atrio J, Schreiber CA, Harvie HS. Cost-effectiveness of Mifepristone Pretreatment for the Medical Management of Nonviable Early Pregnancy: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e201594. doi: 10.1001/jamanetworkopen.2020.1594. PMID 32215633
- [Derived] Clement EG, Horvath S, McAllister A, Koelper NC, Sammel MD, Schreiber CA. The Language of First-Trimester Nonviable Pregnancy: Patient-Reported Preferences and Clarity. Obstet Gynecol. 2019 Jan;133(1):149-154. doi: 10.1097/AOG.0000000000002997. PMID 30531561
- [Derived] Schreiber CA, Creinin MD, Atrio J, Sonalkar S, Ratcliffe SJ, Barnhart KT. Mifepristone Pretreatment for the Medical Management of Early Pregnancy Loss. N Engl J Med. 2018 Jun 7;378(23):2161-2170. doi: 10.1056/NEJMoa1715726. PMID 29874535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We randomly assigned 300 women who had an anembryonic gestation or in whom embryonic or fetal death was confirmed to receive pretreatment with 200 mg of mifepristone, orally, followed by 800 μg of misoprostol, administered vaginally (mifepristone-pretreatment group), or 800 μg of misoprostol alone, administered vaginally (misoprostol-alone group).
Groups:
- Misoprostol: 800 micrograms of vaginal misoprostol alone
  Misoprostol
- Misoprostol Plus Mifepristone: 800 micrograms vaginal misoprostol, preceded by 200 milligrams oral mifepristone 24 hours prior
  Misoprostol
  Mifepristone
Period: Overall Study
Arm/Group | Misoprostol | Misoprostol Plus Mifepristone
Started | 151 | 149
Completed | 149 | 148
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol | Misoprostol Plus Mifepristone | Total
Number analyzed (Participants) | 151 | 149 | 300
Age, Customized [Mean (Full Range); unit: years]
  Participant's age | 30.2 [18 to 46] | 30.7 [18 to 46] | 30.4 [18 to 46]
Sex: Female, Male [Count of Participants; unit: Participants] — Only females where included in this study.
  Participants
    Female | 151 | 149 | 300
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 9 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 67 | 65 | 132
  White | 52 | 57 | 109
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 18 | 39
Region of Enrollment [Number; unit: participants]
  United States | 151 | 149 | 300
Diagnosis [Count of Participants; unit: Participants]
  Anembryonic gestation | 37 | 40 | 77
  Embryonic of fetal death | 114 | 109 | 223

OUTCOME MEASURES:

1. Primary Outcome: Gestational Sac Expulsion With One Treatment Dose on Day 3 (Visit 2) and no Need for Additional Medical or Surgical Intervention Within 30 Days of Treatment.
Time Frame: Day 3 (visit 2) and up to 30 days following visit (to ensure surgical measures were not done
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol | Misoprostol Plus Mifepristone
Number analyzed (Participants) | 149 | 148
Participants | 100 | 124

2. Primary Outcome: Gestational Sac Expulsion by the Second Follow-up Visit at Day 8
Time Frame: Day 8 (visit 3) and up to 30 day to ensure additional measures were not done (surgical)
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol | Misoprostol Plus Mifepristone
Number analyzed (Participants) | 149 | 148
Participants | 111 | 132

3. Primary Outcome: Gestational Sac Expulsion by the 30-day Telephone Call
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol | Misoprostol Plus Mifepristone
Number analyzed (Participants) | 149 | 148
Participants | 113 | 135

4. Primary Outcome: Uterine Asperation
Description: Surgical removal of the miscarriage.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol | Misoprostol Plus Mifepristone
Number analyzed (Participants) | 149 | 148
Participants | 35 | 13

5. Secondary Outcome: Frequency of Serious Adverse Events Between Study Arms.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol | Misoprostol Plus Mifepristone
Number analyzed (Participants) | 151 | 149
Participants | 3 | 5

6. Secondary Outcome: Adverse Event Reported by Participants
Time Frame: 30 Days
Measure: Mean (Full Range); unit: adverse events
Arm/Group | Misoprostol | Misoprostol Plus Mifepristone
Number analyzed (Participants) | 151 | 149
adverse events | 5.6 [0 to 843] | 6.1 [0 to 904]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 30 day time frame
Arm/Group | Misoprostol | Misoprostol Plus Mifepristone
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/149
Serious Adverse Events (participants affected / at risk) | 3/151 | 5/149
Other Adverse Events (participants affected / at risk) | 115/151 | 118/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Misoprostol (N=151) | Misoprostol Plus Mifepristone (N=149)
Bleeding resulting in blood transfusion (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Pelvic Infection (Reproductive system and breast disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Misoprostol (N=151) | Misoprostol Plus Mifepristone (N=149)
Fatigue (General disorders) | 115 | 118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT02012491/Prot_SAP_000.pdf